CLINICAL TRIAL: NCT01178112
Title: Phase I Study of Trientine and Carboplatin in Patients With Advanced Malignancies
Brief Title: Trientine and Carboplatin in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0258; NCI-2012-01787 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-08

CONDITIONS: Advanced Cancers
Keywords: Metastasis; Carboplatin; Trientine; Chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trientine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Trientine + Carboplatin MTD Group (Experimental): Trientine starting dose 750 mg by mouth four times a day, two times with meals and two times without meals for 28 days. Carboplatin maximum tolerated dose found in MTD Dose Escalation Group.
  Interventions: Drug: Trientine; Drug: Carboplatin
- MTD Expansion Group (Experimental): Trientine maximum tolerated dose found in MTD Dose Escalation Group; Carboplatin PK Group A, instead of starting on Day 1 of Cycle 1, starts taking trientine daily beginning on Day 2 of Cycle 1. Trientine PK Group B, 1500 mg of trientine is given once without food on Day 21 of Cycle 1 and once without food after the completion of carboplatin on Day 1 of Cycle 2. Carboplatin maximum tolerated dose found in MTD Dose Escalation Group
  Interventions: Drug: Trientine MTD; Drug: Carboplatin MTD
- Carboplatin PK Expansion Group (Experimental): Trientine maximum tolerated dose found in MTD Dose Escalation Group; Carboplatin PK Group A, instead of starting on Day 1 of Cycle 1, starts taking trientine daily beginning on Day 2 of Cycle 1. Trientine PK Group B, 1500 mg of trientine is given once without food on Day 21 of Cycle 1 and once without food after the completion of carboplatin on Day 1 of Cycle 2. Carboplatin maximum tolerated dose found in MTD Dose Escalation Group. PK testing blood samples of 4 mL at following time points: 0, 30, 60 minutes, 2, 3, 4, 6, and 24 hours.
  Interventions: Drug: Trientine MTD; Drug: Carboplatin MTD; Other: PK Testing
- Trientine PK Expansion Group (Experimental): Trientine maximum tolerated dose found in MTD Dose Escalation Group; Carboplatin PK Group A, instead of starting on Day 1 of Cycle 1, starts taking trientine daily beginning on Day 2 of Cycle 1. Trientine PK Group B, 1500 mg of trientine is given once without food on Day 21 of Cycle 1 and once without food after the completion of carboplatin on Day 1 of Cycle 2. Carboplatin maximum tolerated dose found in MTD Dose Escalation Group. PK testing blood samples of 4 mL at following time points: 0, 30, 60 minutes, 2, 3, 4, 6, and 24 hours.
  Interventions: Drug: Trientine MTD; Drug: Carboplatin MTD; Other: PK Testing

INTERVENTIONS:
Drug: Trientine — Starting dose 750 mg by mouth four times a day, two times with meals and two times without meals for 28 days.
  Arms: Trientine + Carboplatin MTD Group
Drug: Carboplatin — Starting dose area under curve (AUC) 4 by vein over two hours on day 1, and once every 28 days.
  Other Names: Paraplatin
  Arms: Trientine + Carboplatin MTD Group
Drug: Trientine MTD — Maximum tolerated dose found in MTD Dose Escalation Group; Carboplatin PK Group A, instead of starting on Day 1 of Cycle 1, starts taking trientine daily beginning on Day 2 of Cycle 1. Trientine PK Group B, 1500 mg of trientine is given once without food on Day 21 of Cycle 1 and once without food after the completion of carboplatin on Day 1 of Cycle 2.
  Arms: Carboplatin PK Expansion Group; MTD Expansion Group; Trientine PK Expansion Group
Drug: Carboplatin MTD — Maximum tolerated dose found in MTD Dose Escalation Group
  Other Names: Paraplatin
  Arms: Carboplatin PK Expansion Group; MTD Expansion Group; Trientine PK Expansion Group
Other: PK Testing — Blood samples of 4 mL at following time points: 0, 30, 60 minutes, 2, 3, 4, 6, and 24 hours.
  Arms: Carboplatin PK Expansion Group; Trientine PK Expansion Group

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of trientine and carboplatin that can be given to patients with advanced cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Trientine is designed to remove excess copper in the body, which may cause cancer cells to stop growing.

Carboplatin is designed to block the growth of cancer cells by stopping cell division, which may cause the cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of carboplatin based on when you joined this study. Up to 3 dose levels of the carboplatin will be tested.

Three (3) to 6 participants will be enrolled at each dose level of carboplatin. The first group of participants will receive the lowest dose level of carboplatin . Each new group will receive a higher dose of the carboplatin than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found.

The dose level of trientine will be based on your blood levels of copper. These levels may vary from person to person.

Expansion Groups:

Once the highest tolerable dose of the study drug combination is found, there will be two expansion groups, one group of 28 extra participants (Group A) and one group of 14 extra participants (Group B). Group A will receive the study combination at the highest tolerable dose. Group B will receive extra doses of trientine before starting Day 1 of Cycle 1.

Pharmacokinetic (PK) Groups:

In additional the the Expansion Groups, once the highest tolerable dose of the study drug combination is found, there will also be 2 PK groups. PK testing measures the amount of study drug in the body at different time points. There will be 6 participants in each group. These groups will also receive the study combination at the highest tolerable dose. There will be extra blood draws for both groups and the drug administration schedule will be different from the groups described above.

For all participants, your dose of the study drugs may be lowered if you have any intolerable side effects. You will not receive a higher dose than the dose level that you are first assigned.

Study Drug Administration:

Dose Escalation and Expansion Groups:

On Day 1 of each 28-day cycle, you will receive carboplatin by vein over 2 hours.

Starting on Day 1 of Cycle 1, you will begin taking trientine by mouth several times each day. If you are in Expansion Group B, you will receive extra doses of trientine within the 14 days before Day 1 of Cycle 1. Your study doctor will tell you when to take trientine and whether it should be taken with or without food. You will also be told how many pills to take.

PK Groups:

Both groups will take the study drugs as described above.

However, if you are in PK Group A, instead of on Day 1 of Cycle 1, you will start taking trientine daily beginning on Day 2 of Cycle 1.

If you are in PK Group B, on Day 21 of Cycle 1 and Day 1 of Cycle 2 you will not eat for 2 hours before and 2 hours after you take trientine.

Study Visits:

Within 7 days before the first dose of study drug:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked how well you are able to perform the normal activities of daily living (performance status).
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 1/2 tablespoons) will be drawn to measure the levels of ceruloplasmin (copper-carrying protein) copper, and iron in your blood.
* Women who are able to become pregnant must have a negative blood (about 1 teaspoon) pregnancy test.
* If your doctor thinks it is needed, you may have an electrocardiogram (ECG) and/or an echocardiogram (ECHO) to check your heart function. An ECG is a test that measures the electrical activity of the heart

Every week until the doctor decides your are taking the correct dose of trientine:

* Blood (about 1 teaspoon) will be drawn for routine tests.
* Blood (about 2 teaspoons) will be drawn to measure the levels of ceruloplasmin in your blood.

Every week during Cycle 1, blood (about 1 teaspoon) will be drawn for routine tests.

Once each cycle:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If your study doctor thinks it is needed, blood (about 1 tablespoon) will be drawn to measure levels of copper and iron in your blood.
* You will be asked about any side effects you may be having.

At the end of every 2 cycles (Cycles 2, 4, 6, and so on):

* You will have a CT, MRI, PET scan, and/or x-ray to check the status of the disease.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.

PK Groups:

If you are in PK Group A, blood (about 1 teaspoon each time) will be drawn:

* On Day 1 of Cycle 1, blood will be drawn 7 times over the 6 hours after you receive carboplatin.
* On Day 2 of Cycle 1, blood will be drawn 1 time.
* On Day 1 of Cycle 2, blood will be drawn 7 times over the 6 hours after you receive carboplatin.
* On Day 2 of Cycle 2, blood will be drawn 1 time.

If you are in PK Group B, blood (about 1 teaspoon each time) will be drawn:

* On Day 21 of Cycle 1, blood will be drawn 7 times over the 6 hours after your dose of trientine.
* On Day 22 of Cycle 1, will be drawn 1 time.
* On Day 1 of Cycle 2, will be drawn 7 times over the 6 hours after you receive carboplatin.
* On Day 2 of Cycle 2, blood will be drawn 1 time.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

Within 30 days after your last dose of study drugs, you will have an end-of-study visit. At this visit, the following tests and procedures performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked about any side effects you may be experiencing.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.
* If the study doctor thinks it is needed, you will have a chest x-ray, CT, MRI, and/or PET scan to check the status of the disease.

This is an investigational study. Trientine is FDA approved and commercially available for the treatment of Wilson's disease. Trientine is not FDA approved for the treatment of advanced cancer. Carboplatin is FDA approved and commercially available for the treatment of ovarian cancer. The combination of trientine and carboplatin to treat advanced cancer is investigational.

Up to 72 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have an advanced malignancy that has either failed one or more prior therapies, or for whom there is no established standard of care therapy that prolongs survival by at least 3 months.
2. Only in 1 of 3 expansion cohorts, we will plan to enroll 14 subjects with platinum-resistant malignancy. Patient with platinum-resistant malignancy is defined to have had a treatment-free interval of less than 6 months following a platinum-based regimen.
3. Patient of any age and any gender. However, those who are 12 years old or younger will be eligible after consultation with their pediatric physicians regarding dose initiation and modification of trientine.
4. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Patient is willing to comply with study procedures and follow-up examinations.
6. Patient or primary care taker must be informed of the investigational nature of this study and must sign and give written Institutional Review Board (IRB)-approved informed consent in accordance with institutional guidelines.
7. If patient is of childbearing potential, she or he must agree to practice an effective method of birth control prior to study entry, for the duration of study participation, and for 30 days after the last study dose.
8. Patient has adequate organ functions: serum bilirubin </= 2.0 mg/dL; ALT </= 3 x upper limit of normal (ULN), or ALT </= 5 x ULN if the patient has hepatic metastasis; serum creatinine </= 1.5 mg/dL or a calculated creatinine clearance of at least 60 mL/min.
9. Patient has adequate bone marrow reserve: absolute neutrophil count (ANC) >/= 1,500 /ul, Platelet count >/= 100,000 /ul , and Hemoglobin >/= 9.0 g/dL.

Exclusion Criteria:

1. Patient receiving any concurrent chemotherapy.
2. Underlying medical condition that might be aggravated by treatment or that cannot be controlled, such as active, uncontrolled, serious infection and cardiac dysfunction.
3. Medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk.
4. Known anaphylactic or severe hypersensitivity to study drugs or their analogs.
5. Patient has failed to recover from any prior surgery within 4 weeks of study entry.
6. Patient is pregnant or lactating.
7. Patient has had any treatment specific for tumor control within 3 weeks of dosing with investigational drugs and cytotoxic agents, or within 2 weeks of cytotoxic agent given weekly, or within 6 weeks of nitrosoureas or mitomycin C, or within 5 half-lives of biological targeted agents with half-lives and pharmacodynamic effects lasting less than 5 days (that includes, but is not limited to, erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents), or failure to recover from the toxic effect of any of these therapies prior to study entry.
8. Patient has any signs of intestinal obstruction interfering with nutrition.
9. Patient has a known history of central nervous system (CNS) metastasis unless the patient has had treatment with surgery or radiation therapy, and is neurologically stable.
10. Patient is not able to swallow oral medication.
11. Patient has clinical evidence of copper deficiency (i.e. ceruloplasmin level was less than 15 mg/dL or free serum copper level less than 2.2 ug/dL).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Carboplatin with Trientine | 4 weeks
  MTD defined by dose limiting toxicities (DLTs) that occur in the first cycle (4 weeks). DLT defined as treatment-related grade 3 or greater nonhematological toxicity other than nausea, vomiting, or fatigue.

SECONDARY OUTCOMES:
Treatment Response of Maximum Tolerated Dose (MTD) of Carboplatin with Trientine | After 2, 28 day cycles
  Categorization of response based on immune-related response criteria and Response Evaluation Criteria in Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Fu S, Naing A, Fu C, Kuo MT, Kurzrock R. Overcoming platinum resistance through the use of a copper-lowering agent. Mol Cancer Ther. 2012 Jun;11(6):1221-5. doi: 10.1158/1535-7163.MCT-11-0864. Epub 2012 Apr 5. PMID 22491798
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org